CLINICAL TRIAL: NCT07122154
Title: Future Osteoarthritis Treatment (FOOTSTEP) - Free Open Online Course for All
Brief Title: Future Osteoarthritis Treatment - Free Open Online Course for All
Acronym: FOOTSTEP
Status: Not yet recruiting | Type: Observational
Sponsor: Eva Ekvall-Hansson (Other)
Responsible Party: Sponsor-Investigator, Eva Ekvall-Hansson, Professor in physiotherapy, head of research group, Lund University
Organization: Lund University (Other)
Other Study IDs: 2024-03696-01; R-1012802 (Other Grant/Funding Number: The Swedish Rheumatics Association)
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis (OA)
Keywords: Osteoarthritis; Self-management; Participatory design
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OA group: Persons who are diagnosed with osteoarthritis by a healthcare professional, aged 18 years or older, and willing to participate in a series of workshops and provide informed consent.

SUMMARY:
The basic treatment for osteoarthritis is education and information, often provided as so-called osteoarthritis schools. These can be provided either physically at the health center or digitally. The content is similar in all osteoarthritis schools. It is not clear whether today's osteoarthritis schools contain what people with osteoarthritis are asking for in terms of education and information. The purpose of this project is therefore to highlight what people with osteoarthritis want the osteoarthritis school to contain and whether there is a need for other ways of running osteoarthritis schools than today.

Participating in this project means that you will be invited to a focus group with other people who have osteoarthritis. Focus groups will be held at Forum Medicum, Sölvegatan 19 in Lund and will last approximately 1 hour. There will be several different times to choose from. The conversation in the focus group will be recorded.

The project will collect and register information about you. We will collect information about gender, age, in which joint(s) the person has osteoarthritis and how long they have had osteoarthritis, as well as whether they have participated in any osteoarthritis school and if so, what form (physical or digital). The recorded conversation from the focus group will be transcribed.

DETAILED DESCRIPTION:
Background Osteoarthritis (OA) is one of the most prevalent musculoskeletal disorders, affecting between 7% and 65% of populations globally, depending on calculation methods (1). As a chronic condition, OA cannot be cured; thus, treatment focuses on pain management, functional improvement, and self-management strategies. Current guidelines advocate for basic treatment that includes patient education, physical activity, and, when necessary, weight loss (2). The treatment is often given as patient education. Despite that patient education for OA is offered in many countries round the world, it is not clarified if this fundamental treatments is utilized to all patients in need of adequate OA education ref.

Despite national guidelines updated in 2021 recommending that all individuals with OA be offered basic treatment (3), research has shown that participation rates in OA education programs are low (4). For instance, a study from Sweden found that only 40% of patients diagnosed with OA and awaiting surgery had engaged in OA education (5, 6). This raises critical questions about how many patients in primary care are offered such education and the reasons as to why some patients decline to participate.

Furthermore, it remains unclear whether the existing OA education is tailored to meet the diverse needs and preferences of individuals living with OA. Key aspects such as content relevancy and the format of education, whether digital or in-person, have not been adequately addressed. The current educational approach may not align with modern person-centered care principles (7), which prioritizes care that is responsive to individual patient circumstances and preferences.

This lack of alignment suggests a significant gap in the current OA education framework. With OA increasingly affecting younger individuals (8), there is an urgent need to explore contemporary preferences for treatment formats. Although society has become more digitalized, OA education has not evolved accordingly; it still resembles the models developed over 30 years ago. Övergång till nästa stycke, dvs self-management? Changing OA education towards a design that empowers the patient using a participatory discourse has been called upon REferens Self-management is a crucial component of effective OA care, enabling individuals to take an active role in managing their symptoms and improving their quality of life (2). However, for self-management strategies to be effective, they must be grounded in education that is relevant, accessible, and tailored to individual needs (9). When OA care shifts to emphasize person-centered approaches, it is essential to adapt educational formats and content to better meet the needs of individuals with osteoarthritis.

Hence, this study aims to address these gaps by conducting a qualitative study to explore the needs and preferences of individuals with OA regarding support for self-management. By identifying how best to deliver education that resonates with patients' realities, we can enhance their quality of life and ensure that treatment aligns with contemporary expectations for healthcare.

Methods /design Study aims This study aims to explore the knowledge, beliefs, and behaviors of individuals with osteoarthritis, and to identify strategies for encouraging effective use of educational resources to support their self-management.

Study objectives

1. To understand patient's knowledge and beliefs about osteoarthritis
2. To investigate any barriers to using available information about osteoarthritis
3. To identify strategies for encouraging greater engagement with educational recourses and support tools.

Study Design A mixed-method research approach will be employed, combining questionnaires, workshops, and journey mapping to gain a comprehensive understanding of the participants' perspectives and experiences.

Participants Recruitment Strategy: Recruitment of adults >18 years with OA will take place from October 2025 through advertisment on social media. A webpage will be created with information about the project. Links to this page will be posted on Lund University's Facebook, Instagram, LinkedIn and other relevant forums. Participants can access a link to the webpage where they will find the participant information sheet (PIS). The PIS will explain the purpose of the study and its content, clarify the benefits and any risks, who constitutes the research team, that participation is fully voluntary, and that they have the right to cancel participation at any time. All data collected will be encrypted and saved in a secure online repository held by Lund University, with participant data only accessible by the research team.

Inclusion Criteria:

* men and women diagnosed with osteoarthritis by a healthcare professional.
* Aged 18 years or older.
* Willing to participate in a series of workshops and provide informed consent.

Sample Size A total of 2-4 workshops will be held, with 8-10 participants in each workshop. The number of workshops and participants is based on achieving data saturation, ensuring a broad range of perspectives while avoiding redundancy in the data.

Study Procedure

1. Understanding patient's Knowledge and Beliefs About Osteoarthritis

   To capture participants' knowledge and beliefs about osteoarthritis, we will develop a study-specific questionnaire. The questionnaire will include both closed and open-ended questions designed to assess:
   * Baseline knowledge of osteoarthritis
   * Beliefs and attitudes toward osteoarthritis and management of the illness and disease?
   * Understanding of self-management and available resources This method allows for efficient data collection from a large sample and provides insights into patterns and variations in knowledge and beliefs among participants.
2. Understanding Why Available Information Is Not Used

   To investigate any barriers to using available information about osteoarthritis, problem solving techniques (10), will be employed:
   * Journey Mapping: Participants who have engaged with osteoarthritis-related information will map their journey through the system of information. This will involve identifying:

     * Information sources they accessed
     * How they discovered these sources
     * Their perceived usefulness and sufficiency of…
     * Whether and how they applied the strategies suggested
     * Application of strategies suggested in the resources. Participants will rate each step based on ease of access, relevance, and perceived value.
   * Scenario Creation and/or Persona Development: For participants who have not used available resources, hypothetical scenarios and/or personas will be developed to explore potential barriers. These methods provide ethical and creative ways to explore diverse experiences.
3. Encouraging Engagement With Educational Resources

Workshops will use ideation techniques to generate actionable strategies for increasing engagement:

• Brainwriting or Group Passing (11): Participants will engage in a structured brainstorming session using the "Brainwriting" technique. This method involves writing down individual ideas and preferences for osteoarthritis education and support in response to prompts (e.g., "What kind of information would help you manage your osteoarthritis better?"). This allows each participant build on each other's ideas to propose innovative solutions.

Data Collection Audio and Video Recording: Each workshop will be audio and video recorded (with participant consent) to ensure that no valuable insights are lost. These recordings will be transcribed verbatim for analysis.

Field Notes: The moderator and any assistant researchers will take detailed field notes, capturing non-verbal cues, group dynamics, and key points raised during the discussion that may not be fully evident in the transcripts.

Data Analysis The data from the workshops will be analyzed using thematic analysis (12- 14). This involves systematically coding the data to identify patterns, themes, and subthemes related to participant needs, preferences, and experiences.

* Initial coding will be inductive, allowing themes to derive naturally from the data.
* Once preliminary themes have been identified, a second round of coding will be conducted to refine and group related themes into overarching categories.

Validation of Findings: Once the themes have been derived, a summary of the findings will be shared with participants in a follow-up session (or via email if participants prefer) to allow the participants to clarify or expand on their responses. This step is done to ensure that the researchers' interpretations are accurate.

Data management and data protection All data collected within the project will be encrypted and saved in a secure repository held by Lund University, with participant data only accessible by the research team. This refers to the ethics applications/opinions/approvals, recruitment process, personal data collected from participants by any means (paper or digital). Each participant will be given a unique identification number. All identifiable data will be kept in a locked cabinet; and forms with identifiable data will be kept separate from the outcome data. Recordings of qualitative data will be destroyed once transcribed.

Ethical Considerations Informed Consent: All participants will be fully informed about the study's aims, procedures, and their rights as participants. They will provide written consent prior to participation.

Confidentiality: All personal data, including workshop recordings and transcripts, will be securely stored and anonymized to protect participant confidentiality. Only the research team will have access to the raw data, and findings will be presented in a way that does not identify any individual participant.

Ethics Approval: This study will be conducted in accordance the Declaration of Helsinki and Good Clinical Practice Guidelines and is approved by the Swedish Ethical Review Authority.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with osteoarthritis by a healthcare professional.
* Aged 18 years or older.
* Willing to participate in a series of workshops and provide informed consent

Exclusion Criteria:

* Not speaking Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons aged 18 years and above, diagnosed with Osteoarthritis by a healthcare professional, and willing to particpa in a series of workshops
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Experiences | The outcome is collected at one single workshop
  A qualitative research approach will be employed, using workshops as the primary method of data collection. Workshops will allow for dynamic and interactive engagement, where participants can openly share their perspectives, collaborate, and build on each other's ideas.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ekvall Hansson, Professor, Principal Investigator — Lund University, Medical Faculty, Dep of Health Sciences
Locations (1):
- Lund university, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared since sharing is not allowed according to Swedish ethical law.

REFERENCES:
- [Background] Larsson I PhD, PT, Sunden A PhD, PT, Ekvall Hansson E PhD, PT. Persons' various experiences of learning processes in patient education for osteoarthritis, a qualitative phenomenographic approach. Physiother Theory Pract. 2019 Aug;35(8):738-747. doi: 10.1080/09593985.2018.1457111. Epub 2018 Mar 30. PMID 29601226
- [Background] Hagen KB, Smedslund G, Osteras N, Jamtvedt G. Quality of Community-Based Osteoarthritis Care: A Systematic Review and Meta-Analysis. Arthritis Care Res (Hoboken). 2016 Oct;68(10):1443-52. doi: 10.1002/acr.22891. Epub 2016 Sep 16. PMID 26991934
- [Background] Cronstrom A, Nero H, Lohmander LS, Dahlberg LE. On the waiting list for joint replacement for knee osteoarthritis: Are first-line treatment recommendations implemented? Osteoarthr Cartil Open. 2020 Mar 10;2(2):100056. doi: 10.1016/j.ocarto.2020.100056. eCollection 2020 Jun. PMID 36474591
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997
- [Background] Allen KD, Thoma LM, Golightly YM. Epidemiology of osteoarthritis. Osteoarthritis Cartilage. 2022 Feb;30(2):184-195. doi: 10.1016/j.joca.2021.04.020. Epub 2021 Sep 14. PMID 34534661